CLINICAL TRIAL: NCT02589015
Title: Correlation of Neck Circumference With Difficult Mask Ventilation and Difficult Laryngoscopy in Morbidly Obese Turkish Patients: A Prospective Clinical Trial
Brief Title: Correlation of Neck Circumference With Difficult Mask Ventilation and Difficult Laryngoscopy in Morbidly Obese Patients
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Aylin Ozdilek, MD, Istanbul University
Other Study IDs: 02-887/2
Record Dates: First submitted 2015-08-20; First posted 2015-10-28 (Estimated); Last update posted 2016-02-11 (Estimated); Status verified 2016-02

CONDITIONS: Morbid Obesity
Keywords: morbid obesity; neck circumference; difficult mask ventilation; difficult laryngoscopy
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The aim of this study is to determine the correlation of neck circumference with difficult mask ventilation and laryngoscopy in morbidly obese patients.

DETAILED DESCRIPTION:
Patients' Mallampati score, upper lip bite test, neck mobility, teeth abnormalities were evaluated preoperatively. Mouth opening, sternomental and thyromental distances, neck circumference, thoracic circumference, breast circumference , belly circumference and hip circumference were measured preoperatively.

After anesthesia induciton with propofol and rocuronium, patients' mask ventilation difficulty was evaluated as defined below: V1- Ventilated by single anesthesist easily; V2- Ventilated by single anesthesist with oral airway; V3- Ventilated by two anesthesists; V4- Unable to mask ventilate. V3 and V4 was defined as difficult mask ventilation.

Laringoscopy was performed with MacIntosh laryngoscop and Cormack Lehane (CL) score was evaluated. CL score III and IV were defined as difficult laryngoscopy.

ELIGIBILITY:
Inclusion Criteria:

* BMI >= 40
* American Society of Anesthesiologists (ASA) Physical Status I-III
* Patients applied for elective surgery

Exclusion Criteria:

* BMI < 40
* maxillofacial tumor or fracture
* mass at the neck
* mass in the thorax or mediastina
* scar at the neck area
* previous radiotherapy history to neck area
* history of cervical vertebra operations
* cervical vertebra structure abnormality

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with body mass index (BMI) > = 40, applied for elective surgery.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2015-03; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Correlation of difficult laryngoscopy with neck circumference | Cormack Lehane score was assessed during laryngoscopy
  Cormack Lehane scores III and IV were defined as difficult laryngoscopy.
Correlation of difficult mask ventilation with neck circumference | Ventilation difficulty scale was assessed during mask ventilation
  Patients' mask ventilation difficulty was evaluated as defined below: V1- Ventilated by single anesthesist easily; V2- Ventilated by single anesthesist with oral airway; V3- Ventilated by two anesthesists; V4- Unable to mask ventilate. V3 and V4 was defined as difficult mask ventilation.

SECONDARY OUTCOMES:
Correlation of difficult laryngoscopy with modified mallampati score | Cormack Lehane score was assessed during laryngoscopy
  Cormack Lehane scores III and IV were defined as difficult laryngoscopy.
Correlation of difficult mask ventilation with modified mallampati score | Ventilation difficulty scale was assessed after during mask ventilation
  Patients' mask ventilation difficulty was evaluated as defined below: V1- Ventilated by single anesthesist easily; V2- Ventilated by single anesthesist with oral airway; V3- Ventilated by two anesthesists; V4- Unable to mask ventilate. V3 and V4 was defined as difficult mask ventilation.
Correlation of difficult laryngoscopy with neck movement | Cormack Lehane score was assessed during laryngoscopy
  Cormack Lehane scores III and IV were defined as difficult laryngoscopy.
with neck movement | Ventilation difficulty scale was assessed during mask ventilation
  Patients' mask ventilation difficulty was evaluated as defined below: V1- Ventilated by single anesthesist easily; V2- Ventilated by single anesthesist with oral airway; V3- Ventilated by two anesthesists; V4- Unable to mask ventilate. V3 and V4 was defined as difficult mask ventilation.
Correlation of difficult laryngoscopy with dentition | Cormack Lehane score was assessed during laryngoscopy
  Cormack Lehane scores III and IV were defined as difficult laryngoscopy.
Correlation of difficult mask ventilation with dentition | Ventilation difficulty scale was assessed during mask ventilation
  Patients' mask ventilation difficulty was evaluated as defined below: V1- Ventilated by single anesthesist easily; V2- Ventilated by single anesthesist with oral airway; V3- Ventilated by two anesthesists; V4- Unable to mask ventilate. V3 and V4 was defined as difficult mask ventilation.
Correlation of difficult laryngoscopy with upper lip bite test | Cormack Lehane score was assessed during laryngoscopy
  Cormack Lehane scores III and IV were defined as difficult laryngoscopy
Correlation of difficult mask ventilation with upper lip bite test | Ventilation difficulty scale was assessed during mask ventilation
  Patients' mask ventilation difficulty was evaluated as defined below: V1- Ventilated by single anesthesist easily; V2- Ventilated by single anesthesist with oral airway; V3- Ventilated by two anesthesists; V4- Unable to mask ventilate. V3 and V4 was defined as difficult mask ventilation.
Correlation of difficult laryngoscopy with mouth opening | Cormack Lehane score was assessed during laryngoscopy
  Cormack Lehane scores III and IV were defined as difficult laryngoscopy
Correlation of difficult mask ventilation with mouth opening | Ventilation difficulty scale was assessed during mask ventilation
  Patients' mask ventilation difficulty was evaluated as defined below: V1- Ventilated by single anesthesist easily; V2- Ventilated by single anesthesist with oral airway; V3- Ventilated by two anesthesists; V4- Unable to mask ventilate. V3 and V4 was defined as difficult mask ventilation.
Correlation of difficult laryngoscopy with sternomental distance | Cormack Lehane score was assessed during laryngoscopy
  Cormack Lehane scores III and IV were defined as difficult laryngoscopy
Correlation of difficult mask ventilation with sternomental distance | Ventilation difficulty scale was assessed during mask ventilation
  Patients' mask ventilation difficulty was evaluated as defined below: V1- Ventilated by single anesthesist easily; V2- Ventilated by single anesthesist with oral airway; V3- Ventilated by two anesthesists; V4- Unable to mask ventilate. V3 and V4 was defined as difficult mask ventilation.
Correlation of difficult laryngoscopy with breast circumference | Cormack Lehane score was assessed during laryngoscopy
  Cormack Lehane scores III and IV were defined as difficult laryngoscopy
Correlation of difficult mask ventilation with breast circumference | Ventilation difficulty scale was assessed during mask ventilation
  Patients' mask ventilation difficulty was evaluated as defined below: V1- Ventilated by single anesthesist easily; V2- Ventilated by single anesthesist with oral airway; V3- Ventilated by two anesthesists; V4- Unable to mask ventilate. V3 and V4 was defined as difficult mask ventilation.
Correlation of difficult laryngoscopy with thorax circumference | Cormack Lehane score was assessed during laryngoscopy
  Cormack Lehane scores III and IV were defined as difficult laryngoscopy
Correlation of difficult mask ventilation with thorax circumference | Ventilation difficulty scale was assessed during mask ventilation
  Patients' mask ventilation difficulty was evaluated as defined below: V1- Ventilated by single anesthesist easily; V2- Ventilated by single anesthesist with oral airway; V3- Ventilated by two anesthesists; V4- Unable to mask ventilate. V3 and V4 was defined as difficult mask ventilation.
Correlation of difficult laryngoscopy with waist circumference | Cormack Lehane score was assessed during laryngoscopy
  Cormack Lehane scores III and IV were defined as difficult laryngoscopy
Correlation of difficult mask ventilation with waist circumference | Ventilation difficulty scale was assessed during mask ventilation
  Patients' mask ventilation difficulty was evaluated as defined below: V1- Ventilated by single anesthesist easily; V2- Ventilated by single anesthesist with oral airway; V3- Ventilated by two anesthesists; V4- Unable to mask ventilate. V3 and V4 was defined as difficult mask ventilation.
Correlation of difficult laryngoscopy with hip circumference | Cormack Lehane score was assessed during laryngoscopy
  Cormack Lehane scores III and IV were defined as difficult laryngoscopy
Correlation of difficult mask ventilation with hip circumference | Ventilation difficulty scale was assessed during mask ventilation
  Patients' mask ventilation difficulty was evaluated as defined below: V1- Ventilated by single anesthesist easily; V2- Ventilated by single anesthesist with oral airway; V3- Ventilated by two anesthesists; V4- Unable to mask ventilate. V3 and V4 was defined as difficult mask ventilation.

CONTACTS AND LOCATIONS:
Overall Officials: Güniz Köksal, Professor, Study Director — Istanbul University Cerrahpasa Medical Faculty
Locations (1):
- Istanbul University Cerrahpasa Medical Faculty, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ozdilek A, Beyoglu CA, Erbabacan SE, Ekici B, Altindas F, Vehid S, Koksal GM. Correlation of Neck Circumference with Difficult Mask Ventilation and Difficult Laryngoscopy in Morbidly Obese Patients: an Observational Study. Obes Surg. 2018 Sep;28(9):2860-2867. doi: 10.1007/s11695-018-3263-3. PMID 29687341